CLINICAL TRIAL: NCT01751568
Title: Phase I/II Dose-Finding, Safety, Tolerance, and Pharmacokinetics Study of a Raltegravir-Containing Antiretroviral Therapy (ART) Regimen in HIV-Infected and TB Co-Infected Infants and Children
Brief Title: Safety, Tolerance and Pharmacokinetics of Raltegravir-Containing Antiretroviral Therapy in Infants, Children Infected With HIV and TB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1101; 11831 (Registry Identifier: DAIDS-ES Number); IMPAACT P1101
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: ≥ 2 to < 6 years of age on TB treatment (Experimental): Participants in this cohort received chewable raltegravir tablets, starting dose of 12 mg/kg (up to a maximum of 800 mg) orally twice daily, in addition to two NRTIs to treat HIV as part of standard of care, and a rifampicin-containing regimen to treat TB. After a study visit at Day 5 to 8, a fourth ARV medication was added to the regimen.
  Interventions: Drug: Raltegravir
- Cohort 2: ≥ 6 to < 12 years of age on TB treatment (Experimental): Participants in this cohort received chewable raltegravir tablets, starting dose of 12 mg/kg (up to a maximum of 800 mg) orally twice daily, in addition to two NRTIs to treat HIV as part of standard of care, and a rifampicin-containing regimen to treat TB. After a study visit at Day 5 to 8, a fourth ARV medication was added to the regimen.
  Interventions: Drug: Raltegravir
- Cohort 3: : ≥ 4 weeks to < 2 years of age on TB treatment (Experimental): Participants in this cohort received chewable raltegravir tablets (as a dispersible tablet), starting dose of 12 mg/kg (up to a maximum of 800 mg) orally twice daily, in addition to two NRTIs to treat HIV as part of standard of care, and a rifampicin-containing regimen to treat TB. After a study visit at Day 5 to 8, a fourth ARV medication was added to the regimen.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Chewable raltegravir tablets, initially dosed at 12 mg/kg (up to a maximum of 800 mg) orally twice daily.

SUMMARY:
People who are infected with HIV and tuberculosis (TB) need to receive medications that treat both diseases safely and effectively. This study enrolled infants and children infected with HIV and TB and evaluated the safety and tolerance of an antiretroviral (ARV) treatment regimen for HIV that contains raltegravir when administered with a TB treatment regimen that includes rifampicin. Study researchers aimed to determine the most effective dose of raltegravir for infants and children when taken with rifampicin.

DETAILED DESCRIPTION:
People who are infected with HIV are also at risk for becoming infected with TB, particularly in many resource-limited settings, including Sub-Saharan Africa. Rifampicin is a medication commonly used to treat TB. There is a need for HIV treatment regimens that contain newer ARV medications that are well-tolerated and have minimal interactions with rifampicin-containing TB medication regimens. This study enrolled HIV-infected infants and children: who had never taken any ARV medications or who had not received ARVs for at least 30 days prior to study entry; and who were infected with TB and were taking or were starting a TB medication regimen that included rifampicin. The purpose of this study was to evaluate the safety and tolerance of raltegravir-containing ARV regimens to treat HIV when administered with a rifampicin-containing regimen used to treat TB in infants and children. Study researchers also evaluated the pharmacokinetics of the medications (i.e., how medication is absorbed and processed in the body) and determined the most effective dose of raltegravir when administered with a TB regimen that contains rifampicin.

During the study, researchers continuously monitored participant data for safety and other factors. Researchers could adjust the dose of raltegravir given to a group of participants prior to enrolling additional participants.

At study entry, participants underwent a medical and medication history review, physical examination, medication adherence assessment, blood collection, and urine collection. Participants received chewable raltegravir tablets twice daily, and they also took their TB medications, including rifampicin, and two nucleoside reverse transcriptase inhibitor (NRTI) ARV medications chosen by participants' doctors. This study provided raltegravir to participants; all other medications were prescribed by participants' own doctors.

At a study visit at Days 5 to 8, participants remained in the clinic for about 12 hours. They took part in the same study procedures that occurred at the entry visit, but they also had small amounts of blood collected several times throughout the 12 hours to measure the amount of medication in the blood. After the Day 5 to 8 visit, participants began receiving a fourth ARV medication chosen by their doctor, in addition to the other medications. Participants continued receiving raltegravir until they stopped taking their TB medications. They continued to take the third ARV medication and the other two ARV medications for three months after they stopped receiving raltegravir and the TB medications.

Additional study visits occurred at Day 14, Weeks 4 and 8, every 4 weeks until the participant stopped receiving raltegravir and their TB medications, and 4 and 12 weeks after stopping raltegravir and the TB medications. These study visits included the same study procedures that occurred at study entry. Participants were expected to participate in the study for a total of about 4 to 9 months.

Note that out of the forty (40) participants enrolled only (39) participants received the study treatment (raltegravir). The total enrollment for Cohort 1 was thirteen (13) participants, with only twelve (12) who received raltegravir. Therefore, the results of this submission is based on the 39 participants who received raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than or equal to 3.5 kg at entry
* Confirmation of HIV-1 infection was defined as positive results from two samples collected at different time points. All samples tested must be whole blood, serum, or plasma. For studies conducted under an Investigational New Drug (IND), all test methods should be Food and Drug Administration (FDA)-approved if available. If FDA-approved methods are not available, test methods should be verified according to good clinical laboratory practice (GCLP) and approved by the International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) Laboratory Center. More information on this criterion can be found in the protocol.
* ARV treatment naïve or did not received ARVs for at least 30 days prior to entry. Note: Participants with prior exposure to ARVs for prevention of mother-to-child transmission (PMTCT) or treatment - regardless of duration - were eligible provided the participant did not received ARVs for at least 30 days prior to entry. The reasons for interruption could include drug toxicity, poor adherence, or treatment failure that preceded enrollment and was not imposed by study staff. ARVs should not be withheld for the purposes of enrollment into the study and against the participant's best interest.
* ARV treatment eligible as defined by:

  1. Country-specific guidelines OR
  2. World Health Organization (WHO) pediatric treatment algorithm (http://apps.who.int/iris/bitstream/10665/208825/1/9789241549684_eng.pdf?ua=1)
* Diagnosis of pulmonary TB or TB adenitis. More information on this criterion can be found in the protocol.
* Participant initiated at least a 2-drug TB regimen containing rifampicin, and had tolerated at least 1 week of the TB drug regimen prior to initiation of raltegravir. Note: TB treatment was allowed to be started after being diagnosed by the site investigator. Treatment regimens included isoniazid, pyrazinamide, ethambutol and streptomycin in addition to rifampicin. ART ideally started within 2 weeks of starting TB treatment. A patient who had started therapy for TB elsewhere but was not yet been started on ART was eligible for enrollment provided they did not have greater than 20 weeks of TB therapy. Delay between starting TB treatment and ART was not encouraged, and local or international guidelines should be followed for managing TB and HIV coinfection in infants and children.
* Female participant who was of child bearing potential and sexually active agreed to use two reliable methods of contraception, including a medically accepted barrier method of contraception (e.g., female/male condoms, diaphragm or cervical cap with a cream or gel that kills sperm (excluding nonoxydyl-9), intrauterine device [IUD], others) together with another reliable form of contraception while on study and for 4 weeks after stopping raltegravir.
* Parent, legal guardian, or designated guardian according to country-specific guidelines provided signed informed consent and to have the participant followed at the clinical site

Exclusion Criteria:

* Greater than or equal to Grade 2 aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at screening, which must be within 30 days of entry. Note: Participants were allowed to be re-screened provided that they had at least 4 weeks of TB treatment remaining at the time of entry.
* Any greater than or equal to Grade 4 clinical toxicity or laboratory result at screening except fever, chills, fatigue or malaise, unintentional weight loss, and dyspnea or respiratory distress that could be associated with TB
* Acute, serious infections other than TB requiring active treatment (e.g., Pneumocystis jirovecii [previously Pneumocystis carinii] pneumonia [PCP], cryptococcal meningitis, etc.). Infants and children diagnosed with acute bacterial pneumonia at time of diagnosis of TB may be included. Prophylaxis against opportunistic infections was allowed.
* Diagnosis of Kwashiorkor (less than 80% expected weight-for-age with the presence of edema and hypoalbuminemia)
* Current chemotherapy for active malignancy and history of chemotherapy discontinued within 1 year of entry
* Rifampicin therapy of greater than 20 weeks duration immediately prior to enrollment
* Known or suspected multidrug resistant (MDR) or extensively drug resistant (XDR) TB, including contact with a documented MDR or XDR TB source case, as these may require longer duration of therapy or non-rifampicin containing regimen. Note: Participants found to have MDR or XDR TB before or during the study were informed of their illness and referred for appropriate care as determined by local guidelines.
* Current TB regimen containing rifabutin, macrolides, and any other anti-mycobacterial agents with known interactions with raltegravir
* Any clinically significant diseases (other than HIV and TB infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study
* Participant who was pregnant or breastfeeding
* Participant who was unlikely to adhere to the study procedures or keep appointments
* Participant who was planning to relocate during the study to a non-IMPAACT study site
* Participant who was taking any disallowed medications.

Ages: 4 Weeks to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Meyers, MD, Study Chair — Bamboo Grove, Wan Chai, Hong Kong, People's Republic of China; Paul Krogstad, MD, Study Chair — University of California, Los Angeles
Locations (4):
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
  - Famcru Crs, Cape Town, Western Cape

REFERENCES:
- [Background] Lawn SD, Myer L, Bekker LG, Wood R. Burden of tuberculosis in an antiretroviral treatment programme in sub-Saharan Africa: impact on treatment outcomes and implications for tuberculosis control. AIDS. 2006 Aug 1;20(12):1605-12. doi: 10.1097/01.aids.0000238406.93249.cd. PMID 16868441
- [Background] Walters E, Cotton MF, Rabie H, Schaaf HS, Walters LO, Marais BJ. Clinical presentation and outcome of tuberculosis in human immunodeficiency virus infected children on anti-retroviral therapy. BMC Pediatr. 2008 Jan 11;8:1. doi: 10.1186/1471-2431-8-1. PMID 18186944
- [Derived] Krogstad P, Samson P, Acosta EP, Moye J, Townley E, Bradford S, Brown E, Denson K, Graham B, Hovind L, Sise T, Teppler H, Mathiba SR, Fairlie L, Winckler JL, Slade G, Meyers T; International Maternal Pediatric Adolescent AIDS Clinical Trials Network P1101 Team. Pharmacokinetics and Safety of a Raltegravir-Containing Regimen in Children Aged 4 Weeks to 2 Years Living With Human Immunodeficiency Virus and Receiving Rifampin for Tuberculosis. J Pediatric Infect Dis Soc. 2021 Mar 26;10(2):201-204. doi: 10.1093/jpids/piaa039. PMID 32448902
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf?sfvrsn=8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual occurred between November 2014 and April 2019 in four (4) sites from South Africa.
Period: Overall Study
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Started | 13 | 14 | 13
Completed | 12 | 14 | 13
Not Completed | 1 | 0 | 0
Not completed — Participant never started treatment of raltegravir, was taken off-study. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants who enrolled and received raltegravir.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment | Total
Number analyzed (Participants) | 12 | 14 | 13 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.55 [2.95 to 5.55] | 8.55 [7.10 to 10.00] | 1.00 [0.90 to 1.50] | 3.70 [1.50 to 7.20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 17
  Male | 7 | 7 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 14 | 13 | 39
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black Non-Hispanic | 11 | 14 | 13 | 38
  Hispanic (Regardless of Race) | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 12 | 14 | 13 | 39
Log10 RNA [Median (Inter-Quartile Range); unit: log10(copies/ml)] | 4.91 [4.42 to 5.42] | 4.55 [4.21 to 5.09] | 5.13 [5.01 to 5.60] | 4.97 [4.48 to 5.43]
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 559 [389.50 to 1184.50] | 575 [142 to 704] | 1513 [1337 to 2008] | 808 [439 to 1369]
CD4 Percent [Median (Inter-Quartile Range); unit: percentage] | 15.25 [9.30 to 24.35] | 21.35 [6.60 to 25.40] | 16.80 [15.40 to 19.10] | 16.80 [10.60 to 25.10]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 13.60 [11.80 to 16.90] | 21.30 [20.10 to 24.40] | 8.03 [7.00 to 8.56] | 13.80 [8.56 to 20.70]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Permanently Discontinued Treatment Due to Adverse Event(s) of Greater Than or Equal to Grade 3 Deemed at Least Possibly Related to Raltegravir
Description: Number (Frequency) of participants who permanently discontinued raltegravir study treatment due to an adverse event(s) of greater than or equal to Grade 3, deemed at least possibly related to raltergravir.
Time Frame: Measured from the first dose of raltegravir through the participant's last study visit (median of 34 weeks)
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
Participants | 0 | 1 | 0

2. Primary Outcome: Number of Participants Who Experienced Death, Grade 4 Life-threatening Adverse Events Deemed at Least Possibly Related to Raltegravir
Description: Number (Frequency) of participants who experienced Death, Grade 4 life-threatening adverse events deemed at least possibly related to raltegravir
Time Frame: Measured from the first dose of raltegravir through a participant's last study visit (median of 34 weeks)
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced Grade 4 Non-life Threatening Adverse Event(s) Deemed as Probably or Definitely Related to Raltegravir
Description: Number (Frequency) of Participants who experienced Grade 4 non-life threatening adverse event(s) deemed as probably or definitely related to raltegravir
Time Frame: Measured from the first dose of raltegravir through a participant's last study visit (median of 34 weeks)
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced Adverse Event(s) of Greater Than or Equal to Grade 3 Deemed at Least Possibly Related to Raltegravir
Description: Number (Frequency) of Participants who experienced Adverse event(s) of greater than or equal to Grade 3 deemed at least possibly related to raltegravir
Time Frame: Measured from the first dose of raltegravir through a participant's last study visit (median of 34 weeks)
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
Participants | 1 | 1 | 0

5. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Curve (AUC12h)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (Phoenix WinNonlin 8.1, Certara, Princeton, New Jersey). AUC12h (area-under-the-curve from 0 to 12 hours) were determined using the linear-log trapezoidal rule. Geometric Means (GM) for AUC12h were calculated for each cohort.
Time Frame: At the study visit between days 5 and 8 of raltegravir initiation; A (0.5) mL of blood sample was drawn at each time point: pre-dose (0), 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post dosing.
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose in each Age Cohort
Measure: Geometric Mean (Full Range); unit: h*mg/L
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
h*mg/L | 12.8 [4.0 to 25.8] | 17.2 [10.1 to 31.3] | 14.6 [6.4 to 29.7]

6. Primary Outcome: Pharmacokinetic (PK) Parameter: Concentration at 12h (C12)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (Phoenix WinNonlin 8.1, Certara, Princeton, New Jersey). AUC12h (area-under-the-curve from 0 to 12 hours) were determined using the linear-log trapezoidal rule. Geometric Means (GM) for C12 were calculated for each cohort.
Time Frame: as for outcome 5
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose in each Age Cohort
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
ng/mL | 101.8 [18.8 to 334.9] | 101.2 [48.3 to 354.6] | 47.3 [19.6 to 131.4]

7. Secondary Outcome: Number of Participants Who Failed to Respond Virologically at Week 8, Which Means Having HIV RNA (Copies/mL) Greater Than 400 Copies/mL AND Less Than 1-log10 Drop From Baseline
Description: Number (Frequency) of Participants who failed to respond virologically at Week 8, which includes HIV RNA (copies/mL) greater than 400 copies/mL AND less than 1-log10 drop from baseline. Please note that the protocol definition of virologic response was: achieving at least a 1-log10 reduction from baseline in HIV-1 RNA (copies/mL) or HIV-1 RNA ≤ 400 copies/mL at week 8. An As-Treated (AT) analysis was carried out, such that participants who permanently discontinued treatment before week 8, without evaluable data were not included in the analyses.
Time Frame: Measured at Week 8
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort. Please note that an as-Treated (AT) analysis was carried out, such that participants who permanently discontinued treatment before week 8, without evaluable data were not included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 12 | 12
Participants | 1 | 1 | 1

8. Secondary Outcome: Number of Participants Who Developed of New Opportunistic Infection(s) (OIs)
Description: Number (Frequency) of participants who developed of new opportunistic infection(s) (OIs)
Time Frame: Measured from the first dose of raltegravir through a participant's last study visit (median of 34 weeks)
Population: Includes all participants who received at least one dose of raltegravir at the final recommended dose for the cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
Number analyzed (Participants) | 12 | 14 | 13
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Measured from the first dose of raltegravir through the participant's last study visit (up to 64 weeks).
Description: All new diagnoses, signs/symptoms and laboratory events of ≥Grade 1 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade, were collected. Adverse events (AE) were graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014.
Arm/Group | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 8/12 | 5/14 | 5/13
Other Adverse Events (participants affected / at risk) | 12/12 | 14/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment (N=12) | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment (N=14) | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment (N=13)
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Amylase increased (Investigations) | 2 | 0 | 2
Bilirubin conjugated increased (Investigations) | 2 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 3 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ≥ 2 to < 6 Years of Age on TB Treatment (N=12) | Cohort 2: ≥ 6 to < 12 Years of Age on TB Treatment (N=14) | Cohort 3: : ≥ 4 Weeks to < 2 Years of Age on TB Treatment (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Noninfective myringitis (Ear and labyrinth disorders) | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 4
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Lip erythema (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
Chest pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 1
Acarodermatitis (Infections and infestations) | 1 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1
Body tinea (Infections and infestations) | 1 | 3 | 1
Candida nappy rash (Infections and infestations) | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Gianotti-Crosti syndrome (Infections and infestations) | 0 | 1 | 0
Helminthic infection (Infections and infestations) | 1 | 0 | 0
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 2 | 4 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Varicella (Infections and infestations) | 1 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 5 | 7
Amylase increased (Investigations) | 9 | 11 | 10
Aspartate aminotransferase increased (Investigations) | 6 | 8 | 5
Bilirubin conjugated increased (Investigations) | 1 | 0 | 5
Blood albumin decreased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 4
Blood bicarbonate decreased (Investigations) | 11 | 12 | 12
Blood bilirubin abnormal (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood calcium decreased (Investigations) | 3 | 2 | 1
Blood calcium increased (Investigations) | 1 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 2
Blood glucose decreased (Investigations) | 7 | 8 | 5
Blood glucose increased (Investigations) | 2 | 1 | 2
Blood magnesium decreased (Investigations) | 3 | 5 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 1
Blood potassium increased (Investigations) | 1 | 1 | 9
Blood pressure diastolic increased (Investigations) | 1 | 1 | 1
Blood pressure systolic increased (Investigations) | 1 | 0 | 1
Blood sodium decreased (Investigations) | 11 | 7 | 9
Breath sounds abnormal (Investigations) | 2 | 2 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 11 | 6 | 11
International normalised ratio increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 2 | 6
Neutrophil count decreased (Investigations) | 3 | 5 | 5
Platelet count decreased (Investigations) | 0 | 1 | 2
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pica (Psychiatric disorders) | 0 | 1 | 0
Renal salt-wasting syndrome (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights".

DOCUMENTS (6):
  • Study Protocol: Version 3.0 (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/Prot_003.pdf
  • Study Protocol: Letter of Amendment 1 (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/Prot_004.pdf
  • Study Protocol: Letter of Amendment 2 (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/Prot_005.pdf
  • Statistical Analysis Plan: Primary Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/SAP_001.pdf
  • Statistical Analysis Plan: Pharmacokinetic Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/SAP_002.pdf
  • Informed Consent Form (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT01751568/ICF_000.pdf